CLINICAL TRIAL: NCT02010034
Title: Compassionate Use of Omegaven in the Treatment of Parenteral Nutrition Induced Hepatic Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Medical Center Dallas (Other)
Responsible Party: Principal Investigator, Nandini Channabasappa, MD, Director, Intestinal Rehabilitation Program, Children's Medical Center Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 112010-159
Record Dates: First submitted 2013-08-19; First posted 2013-12-12 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Liver Disease; Impaired Liver Function; Parenteral Nutrition Associated Liver Disease
Keywords: TPN; Liver Function; parenteral nutritional fat emulsions
MeSH Terms: conditions — Liver Diseases | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Compassionate use (Other): This lipid preparation is only being used for compassionate use.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Omegaven will be used in place of soy oil Intralipid

SUMMARY:
This study is being done to determine if an investigational study drug called Omegaven can help to improve liver disease thought to be caused by Total Parenteral Nutrition (TPN). TPN is intravenous feeding (IV feeding tube) that provides patients the nutrients when they are unable to drink fluid or eat food by mouth.

DETAILED DESCRIPTION:
PAtients with direct bilirubin >2gm/dL and short bowel syndrome are eligible for enrollment. Omegaven at 1gm/kg/day will be administered via central venous line instead of standard lipid preparations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 2 months -10 years of age
2. Patients who are PN dependent (unable to meet nutritional needs solely by enteral nutrition) and are expected to require PN for at least another 30 days
3. Patients considered eligible for study participation must have parenteral nutrition associated liver disease (PNALD) as defined by a direct bilirubin of >2.0mg/dL. Other causes of liver disease should be excluded. A liver biopsy is not necessary for treatment
4. 2 consecutive direct bilirubin test results >2.0mg/dl
5. The patient must have failed standard therapies to prevent the progression of liver disease such as surgical treatment, cyclic TPN, avoiding overfeeding, reduction/removal of copper and manganese from TPN, advancement of enteral feeding, and use of ursodiol (Actigall)
6. Subjects who are currently under treatment for PNALD with Compassionate Use Omegaven and have a direct Bilirubin of< 2, but who remain TPN dependent and require continued therapy with Omegaven

Exclusion Criteria:

1. Other known causes of chronic liver disease (hepatitis C, cystic fibrosis, biliary atresia and alpha 1 anti-trypsin deficiency)
2. Enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
3. The parent, guardian, or child is unwilling to provide consent or assent
4. Allergy to any fish product, egg protein, and/or previous allergy to Omegaven
5. Active coagulopathies characterized by on-going bleeding or by a requirement for clotting factor replacement such as fresh frozen plasma or cryoprecipitate to maintain homeostasis
6. Impaired lipid metabolism or severe hyperlipidemia with or without pancreatitis
7. Unstable diabetes mellitus
8. Stroke/embolism
9. Collapse and shock
10. Undefined coma status
11. Active infection at time of initiation of Omegaven® up until such time as child is afebrile with stable vital signs and one negative 48 hour culture

Ages: 2 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2013-08; Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Bilirubin in mg/dL | 12 weeks
  PN associated liver disease can be reversed or its progression halted by using a parenteral fat emulsion prepared from fish oil as measured by normalization of serum levels of hepatic enzymes and bilirubin
  1. after reaching bilirubin levels >2mg/dl, subjects receiving Omegaven will reach a bilirubin level < 2mg/dL faster that patients receiving conventional fat emulsions.

SECONDARY OUTCOMES:
Number of participants with adverse events | 12 weeks
  a. After starting Omegaven on PN, the rate of fatty acid deficiencies and imbalances will be as low as before Omegaven. Also, the rate of triglyceride events >400mg/dL with Omegaven will be similar to that seen with PN administration with soy oil Intralipid.
  B. PN containing Omegaven will be safe for patients with respect to the risk of unexpected bleeding, coagulopathies, and other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Nandini Channabasappa, MD, Principal Investigator — Childrens Health
Locations (1):
- Children's Medical Center of Dallas, Dallas, Texas, United States